CLINICAL TRIAL: NCT05835778
Title: Specific Use-results Study of IMFINZI Intravenous Infusion 120 mg,500mg in Patients With Curatively Unresectable Biliary Tract Cancer
Brief Title: Imfinzi BTC Japan PMS_Japan Post-Marketing Surveillance (PMS) Study - CEI/SCEI
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D933AC00005
Record Dates: First submitted 2023-04-06; First posted 2023-04-28 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

SUMMARY:
To investigate onset of adverse drug reactions in patients with curatively unresectable biliary tract cancer who receive IMFINZI in combination with gemcitabine hydrochloride and cisplatin under actual use in the post-marketing setting.

DETAILED DESCRIPTION:
This investigation will be conducted to investigate onset of adverse drug reactions in patients with curatively unresectable biliary tract cancer who receive IMFINZI Intravenous Infusion 120mg, 500mg in combination with gemcitabine hydrochloride and cisplatin under actual use in the post-marketing setting.

The investigation will be conducted as one of the additional pharmacovigilance activities in the Japan Risk Management Plan of IMFINZI in compliance with the Ministerial Ordinance on Good Post-marketing Study Practice (GPSP Ordinance) and for the purpose of application for reexamination under Article 14-4 of the Act on Securing Quality, Efficacy and Safety of Products Including Pharmaceuticals and Medical Devices.

Among the safety specifications defined in the Japan Risk Management Plan of IMFINZI, the following items are set as the safety specifications for this study.

Interstitial lung disease, Colitis/Severe diarrhoea, Hepatic function disorder/Hepatis/Cholangitis Sclerosing, Endocrine disorders (Dysfunction thyroid, Dysfunction adrenal, Pituitary dysfunction), Type 1 diabetes mellitus, Renal disorder (interstitial nephritis, etc), Myositis, Myocarditis, Myasthenia gravis, Immune thrombocytopenic purpura, Encephalitis, Severe skin disorder, Nerve disorder (including guillain-barre syndrome), Infusion reaction, Pancreatitis, Gastrointestinal perforation, Rhabdomyolysis, Meningitis, Febrile neutropenia during combination treatment with chemotherapy, Embryo-fetal toxicity and Use in patients with a history of organ transplant (including haematopoietic stem cell transplant).

ELIGIBILITY:
Inclusion Criteria:

* Patients with curatively unresectable biliary tract cancer who receive IMFINZI for the first time in combination with gemcitabine hydrochloride and cisplatin.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with curatively unresectable biliary tract cancer
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2025-11-21 (Actual); Study Completion 2025-11-21 (Actual)

PRIMARY OUTCOMES:
Incidence of ADRs | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Toshimitsu Tokimoto, Study Director — AstraZeneca KK
Locations (24):
- Japan (24):
  - Research Site, Aichi
  - Research Site, Aomori
  - Research Site, Chiba
  - Research Site, Ehime
  - Research Site, Fukushima
  - Research Site, Hokkaido
  - Research Site, Hyōgo
  - Research Site, Kagawa
  - Research Site, Kanagawa
  - Research Site, Kyoto
  - Research Site, Miyagi
  - Research Site, Nagano
  - Research Site, Nagasaki
  - Research Site, Nara
  - Research Site, Numakunai
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Saitama
  - Research Site, Shiga
  - Research Site, Shimane
  - Research Site, Shizuoka
  - Research Site, Tochigi
  - Research Site, Tokyo
  - Research Site, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home